CLINICAL TRIAL: NCT03649386
Title: Effect of Heated-humidified Circuit on Arterial Oxygenation in Patients Undergoing One-lung Ventilation for Thoracoscopic Surgery
Brief Title: Heated Circuit for One-lung Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Hyun-Chang Kim, Assistant professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HeatOLV
Record Dates: First submitted 2018-08-22; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: One-lung Ventilation; Oxygenation; Temperature

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Heated breathing circuit will turned off.
  Interventions: Device: Heated and humidified breathing circuit off
- Heat (Experimental): Heated breathing circuit will be turned on.
  Interventions: Device: Heated and humidified breathing circuit on

INTERVENTIONS:
Device: Heated and humidified breathing circuit on — Heated and humidified breathing circuit will be turned on.
  Arms: Heat
Device: Heated and humidified breathing circuit off — Heated and humidified breathing circuit will be turned off.
  Arms: Control

SUMMARY:
One-lung ventilation interrupts oxygenation. The effect of heated humidifed breathing circuit on arterial oxygenation during one-lung ventilation has not been investigated. The investigators will investigate the effect of the heated humidifed breathing circuit on oxygenation during one-lung ventilation in patients undergoing thoracoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist class I-II
* Patients scheduled for one-lung ventilation for thoracoscopic surgery

Exclusion Criteria:

* Obesity
* Severe obstructive or restrictive lung disease
* Preoperative oxygen supply
* Preoperative intubated state or under mechanical ventilatory support
* Baseline arterial partial pressure of oxygen (PaO2) < 70 mmHg
* Symptomatic coronary or peripheral arterial disease
* Renal failure
* Preoperative continuous infusion of inotropes or vasopressor
* Pregnancy

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Arterial oxygenation | At 30 minutes after one-lung ventilation
  Arterial oxygenation (mmHg) will be measured by arterial blood analysis.

SECONDARY OUTCOMES:
Arterial oxygenation | At 0, 15, 45, and 60 minutes after one-lung ventilation
  Arterial oxygenation (mmHg) will be measured by arterial blood analysis.
Mean arterial pressure | At 0, 15, 30, 45, and 60 minutes after one-lung ventilation
  Mean arterial pressure (mmHg) will be measured.
Heart rate | At 0, 15, 30, 45, and 60 minutes after one-lung ventilation
  Heart rate (beats/min) will be measured.
Temperature | At 0, 15, 30, 45, and 60 minutes after one-lung ventilation
  Body temperature (°C) will be measured.
Central venous pressure | At 0, 15, 30, 45, and 60 minutes after one-lung ventilation
  Mean central venous pressure (mmHg) will be measured by a central venous catheter.
Cardiac index | At 0, 15, 30, 45, and 60 minutes after one-lung ventilation
  Cardiac index (l/min/m^2) will be measured by pulse-contour analysis.
Pressure peak | At 0, 15, 30, 45, and 60 minutes after one-lung ventilation
  Peak pressure of ventilation (cmH2O) will be measured.
Pressure plateau | At 0, 15, 30, 45, and 60 minutes after one-lung ventilation
  Plateau pressure of ventilation (cmH2O) will be measured.
Arterial carbon dioxide | At 0, 15, 30, 45, and 60 minutes after one-lung ventilation
  Arterial carbon dioxide will be measured.
Arterial blood acidosis | At 0, 15, 30, 45, and 60 minutes after one-lung ventilation
  Arterial blood acidosis will be measured.
Oxygen saturation of arterial blood | At 0, 15, 30, 45, and 60 minutes after one-lung ventilation
  Oxygen saturation of arterial blood (%) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Chang Kim, MD PhD, Principal Investigator — Keimyung University

IPD SHARING:
Plan to Share IPD: Undecided